CLINICAL TRIAL: NCT03125980
Title: Perioperative CapeOX Chemotherapy Versus Postoperative Chemotherapy for Locally Advanced Resectable Colon Cancer: An Open Label Randomized Controlled Phase III Trial
Brief Title: Perioperative Versus Postoperative CapOX Chemotherapy for Locally Advanced Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Sanjun Cai, Professor, Chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CapeOXcc
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Locally Advanced Colon Cancer
MeSH Terms: interventions — Capecitabine; Postoperative Period

STUDY DESIGN:
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative chemotherapy with CapOX regimen (Experimental)
  Interventions: Drug: capecitabine plus oxaliplatin before and after surgery
- Postoperative chemotherapy with CapOX regimen (Active Comparator)
  Interventions: Drug: capecitabine plus oxaliplatin after surgery

INTERVENTIONS:
Drug: capecitabine plus oxaliplatin before and after surgery — Subjects will receive systemic CapeOX chemotherapy both before and after the radical surgery for at most 4 cycles respectively. They shall have rest after the surgery for at least four weeks before the post-operative chemotherapy. CapOX regimen will be administered as follows:
  1. Oxaliplatin 130 mg/m2 iv continue for 2 hours.D1
  2. Capecitabine 1000mg/m2/d PO Bid,once every morning and evening D1-14
  3. Repeat every 3 weeks (Q3W)
  Arms: Perioperative chemotherapy with CapOX regimen
Drug: capecitabine plus oxaliplatin after surgery — Subjects will first receive radical surgery, then have rest for at least four weeks. Thereafter, subjects will receive systemic CapeOX chemotherapy for at most 8 cycles. CapOX regimen will be administered as follows:
  1. Oxaliplatin 130 mg/m2 iv continue for 2 hours.D1
  2. Capecitabine 1000mg/m2/d PO Bid,once every morning and evening D1-14
  3. Q3W
  Arms: Postoperative chemotherapy with CapOX regimen

SUMMARY:
Adjuvant chemotherapy has been widely adopted worldwide for locally advanced colon cancer. However, more and more studies have found better efficacy and potential advantages of perioperative or neoadjuvant chemotherapy. The sooner the systemic chemotherapy is received, the better suppression it has on activity of tumor growth factors. Pre-operative chemotherapy may eliminate tiny metastases. It may also shrink the invasion of tumor before surgery, and thus reducing operational trauma and expediting recovery. With advances in radiology and tomography, staging before surgery is accurate enough to identify risks and prognosis for patients. The phase II trial conducted by our department has yielded encouraging results (N=47, CapeOX regimen, clinicaltrials.gov NCT02415829): after the neoadjuvant chemotherapy, no subject had disease progression, 68.1% subjects reached complete or partial response. Besides, the toxicity of neoadjuvant CapeOX chemotherapy was acceptable. The present randomized controlled phase III trial will be conducted to further compare efficacy and safety of the neoadjuvant and adjuvant CapeOX chemotherapy for patients with locally advanced resectable colon cancer in China. This study may have two periods, each will last for approximately 5 years. After the first period (n=994), if the results of the test group are better than the control group, the study will be terminated. Otherwise, the study will enter into period 2 (n=376) through selecting out genetically sensitive subjects and repeating the same trial process as period 1.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2;
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment: Neutrophil count≥1.5×109/L, Platelet count≥100×109/L, Hemoglobin≥80g/L, Serum bilirubin≤24umol/L, Alanine aminotransferase and aspartate aminotransferase ≤ 60×IU/L, Serum creatinine≤110 umol/L;
* No current pregnancy or breast-feeding, and subjects at childbearing age shall take method of contraception ;
* Be in a condition to receive a surgery/procedure;
* No second tumor at present or in the past 5 years, except skin basal cell carcinoma, skin squamous cell carcinoma, or any in situ cancer;
* No previous systemic chemotherapy for treating colon cancer;
* No other chemotherapy at the same time;
* Expected lifetime longer than three months;
* Be willing and able to understand the study and to provide written informed consent.

Exclusion Criteria:

* End-stage cachexia patients;
* Cardiopulmonary dysfunction or liver and kidney dysfunction, and unable to tolerate CapeOX chemotherapy;
* Metastatic carcinoma;
* Moderate or above anemia caused by serious local tumor bleeding;
* Incomplete or complete intestinal obstruction;
* Known to be allergic to oxaliplatin or capecitabine;
* Active hepatitis, severe coagulation disorder patients;
* Pregnant or lactating women; or women who have fertility but have not taken at taken adequate contraceptive measures;
* Known to have deficient dihydropyrimidine dehydrogenase (DPD)；
* Have vital organ failure or other severe diseases, including but not limited to coronary heart disease, cardiovascular diseases, or myocardial infarction within 12 months before being included; severe neurological or psychiatric history；severe infection; active disseminated intravascular coagulation;
* Unable or unwilling to abide by the study plan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1370 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 years
  Defined as the length of time from the date of randomization until the first documented date of progression or death from any cause, whichever comes first

SECONDARY OUTCOMES:
R0 resection rate | From the date of randomization until the date of the last patient receiving surgery, assessed up to 40 months
  Defined as the rate of patients whose tumors are completely resected with all the margins being negative
Post-operative TRG staging | From the date of randomization until the date of the last patients receiving surgery, assessed up to 40 months
  Defined as the TRG staging of tumor after surgery
Overall survival (OS) | 5 years
  Defined as the length of time from randomization date until the date of death from any cause
Relapse-free survival (RFS) | 5 years
  Defined as the length of time from the date of randomization until the first documented date of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Xu, M.D, Study Director — Department of Colorectal Surgery Fudan University Shanghai Cancer Center
Locations (1):
- Department of Colorectal Surgery Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Liu F, Tong T, Huang D, Yuan W, Li D, Lin J, Cai S, Xu Y, Chen W, Sun Y, Zhuang J. CapeOX perioperative chemotherapy versus postoperative chemotherapy for locally advanced resectable colon cancer: protocol for a two-period randomised controlled phase III trial. BMJ Open. 2019 Jan 29;9(1):e017637. doi: 10.1136/bmjopen-2017-017637. PMID 30700474